CLINICAL TRIAL: NCT05509595
Title: A Phase 2 Study of Burosumab for Fibroblast Growth Factor-23 Mediated Hypophosphatemia in Fibrous Dysplasia
Brief Title: Burosumab for Fibroblast Growth Factor-23 Mediated Hypophosphatemia in Fibrous Dysplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000798; 000798-D
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01-15

CONDITIONS: Fibrous Dysplasia Of Bone
Keywords: McCune-Albright Syndrome; Rickets; Osteomalacia; Metabolic Bone Disorders
MeSH Terms: conditions — Fibrous Dysplasia of Bone; Fibrous Dysplasia, Polyostotic; Rickets; Osteomalacia; Bone Diseases, Metabolic | interventions — burosumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with burosumab (Experimental): Participants with Fibrous dysplasia/McCune-Albright syndrome (FD/MAS) and hypophosphatemia receive burosumab subcutaneously dosed to the nearest 10mg. Pediatric participants receive 0.8mg/kg subcutaneously every two weeks for 48 weeks. Adult participants receive 0.5mg/kg subcutaneously every four weeks, with the option to receive dose every two weeks, for 48 weeks. All participants receive a minimum dose of 10mg/dose and a maximum of 90mg/dose.
  Interventions: Drug: Burosumab

INTERVENTIONS:
Drug: Burosumab — Human recombinant monoclonal antibody to fibroblast growth factor-23 (FGF23)

SUMMARY:
Background:

Fibrous dysplasia (FD) is a disorder that affects bone growth. Affected bone tissue is weakened, and people with FD are prone to deformities, fractures, and other problems. People with FD may also have low blood phosphate levels. This can make bones even weaker. Better treatments are needed.

Objective:

To test a study drug (burosumab) in people with FD who have low blood phosphate levels.

Eligibility:

People aged 1 year or older who have FD and low blood phosphate levels.

Design:

Participants will visit the NIH 3 times in 48 weeks. Each visit will last 5 to 7 days.

Participants will self-inject burosumab under the skin in their belly, upper arm, or thigh. They (or a caregiver) will do this at home 1 or 2 times a month. They will be trained in person on how to inject the drug. Home injections will be guided via telehealth.

During NIH visits, participants will have a physical exam with blood and urine tests. They will have x-rays of different parts of their body. They will have a radioactive tracer injected into their vein; then they will have a bone scan. They will have tests to assess their strength, walking, and movement. They will complete questionnaires about their pain, mobility, and fatigue levels.

Adult participants may have bone biopsies. These will be done under anesthesia with sedation. Small samples of FD-affected bone will be removed for study.

Between NIH visits, participants will go to a local laboratory for blood and urine tests.

Child participants will have an additional follow-up visit 2 weeks after the final NIH visit.

DETAILED DESCRIPTION:
Study Description:

This will be a phase 2, open-label, single-arm study to evaluate the safety and efficacy of burosumab to normalize serum phosphate levels in subjects with fibrous dysplasia (FD) and fibroblast growth factor 23 (FGF23)-mediated hypophosphatemia.

Objectives:

Primary Objective:

-Evaluate the efficacy of burosumab to normalize serum phosphate levels in subjects with FD and FGF23-mediated hypophosphatemia at 48 weeks.

Secondary Objectives:

* Evaluate the efficacy of burosumab to normalize serum phosphate levels in subjects with FD and FGF23-mediated hypophosphatemia at 24 weeks.
* Evaluate the safety and tolerability of burosumab in patients with FD.
* Evaluate the effect of burosumab on increasing serum phosphate and additional mineral markers.
* Evaluate the impact of burosumab on FD lesion activity.
* Evaluate the effect of burosumab on functional parameters.
* Evaluate the effect of burosumab on pain and health-related quality of life.

Endpoints:

Primary Endpoint:

-The proportion of subjects achieving serum phosphate levels within the target range (Z-score -1 to +2) at Week 48.

Secondary Endpoints:

* Proportion of subjects achieving serum phosphate levels within the target range (Z-score -1 to +2) at Week 24.
* Adverse events and clinical safety laboratory tests for up to 4 weeks after the final burosumab dose (48 weeks for adult subjects, 50 weeks for pediatric subjects).
* Change and percent change from baseline to post-baseline visits in serum phosphate, serum 1,25(OH)2D, ratio of renal tubular maximum reabsorption rate of phosphate to glomerular filtration rate (TmP/GFR).
* Change in FD lesion activity using Fluorine-18 Sodium Fluoride Positron Emission Tomography/Computed Tomography (18F-NaF PET/CT) total lesion activity from baseline to 48 weeks
* Change and percent change in serum bone turnover markers, including procollagen 1 N-terminal propeptide (P1NP), beta crosslaps C-telopeptides (CTX), osteocalcin, and bone-specific alkaline phosphatase from baseline to 48 weeks.
* Change in FD lesion histology and cell proliferation as assessed by minimally invasive bone biopsies from baseline to 48 weeks (adults with capacity to consent only) from baseline to 48 weeks
* Skeletal changes assessed on skeletal survey at baseline and 48 weeks
* Change from baseline to 48 weeks in:

  * Muscle strength
  * Range-of-motion
  * Walking speed (9-minute walk)

Change from baseline to 48 weeks in patient reported outcomes measures:

* Short Form Health Survey 36 (SF-36): adults
* Short Form Health Survey 10 (SF-10): children
* Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity: Pediatric and Parent Proxy version 1.0, Adult version 2.0
* PROMIS Pain Interference: Pediatric and Parent Proxy v 2.0, Adult v 1.1
* PROMIS Mobility: Pediatric and Parent Proxy version 2.0, Adult Mobility Lower Extremity v 1.0
* PROMIS Fatigue: Pediatric and Parent Proxy v 2.0, Adult FACIT 13a v1.0
* Activities of Daily Living Questions: adults and children

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Confirmed diagnosis of fibrous dysplasia
* Serum phosphate <10th percentile for age and sex, AND intact serum FGF23 >=30 pg/mL
* Age >=1 year
* Provision of signed and dated informed consent/assent form
* Stated willingness of subject or Legally Authorized Representative (LAR) to comply with all study procedures and availability for the duration of the study
* For females of reproductive potential: agreement to use highly effective contraception for during study participation. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the participant). Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment.
  * Male sterilization (at least 6 months prior to screening). For female participants on the study the vasectomized male partner should be the sole partner for that participant.
  * Combination of the following (a+b or a+c, or b+c):

    * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
* For males of reproductive potential: use of condoms or other methods described above to ensure effective contraception with partner
* Minimum body weight of 7.5 kilograms

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnancy or lactation
* Known allergic reactions to burosumab or drug component
* Treatment with another investigational drug within 30 days of screening
* Treatment with burosumab within 30 days of screening
* Have any condition which in the opinion of the PI could present a concern for subject safety or difficulty with data interpretation
* Severe renal impairment or end stage renal disease, defined as: pediatric patients with estimated glomerular filtration rate (eGFR) 15 mL/min/1.73m2 to 29 mL/min/1.73m2 or end stage renal disease (eGFR < 15 mL/min/1.73m2), adult patients with creatinine clearance (CLcr) 15 mL/min to 29 mL/min or end stage renal disease (CLcr < 15 mL/min)

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Boyce, M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and the Clinical Trials Registration and Results Information Submission rule.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Results from this trial will be made available 12 months after the primary study completion date
Access Criteria: Investigators from NIH and Ultragenyx and Kyowa Kirin will consider requests from qualified researchers for access to clinical data.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000798-D.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With Burosumab
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment With Burosumab: Participants treated with burosumab
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Serum Phosphate Levels Within the Target Range at Week 48
Description: The proportion of participants who achieved serum phosphate levels within the target range (Z-score -1 to +2) at week 48. Analysis was done by dividing the number of number of participants who achieved serum level by the number of participants analyzed.
Time Frame: Week 48
Population: Modified intent to treat population
Measure: Number; unit: Proportion of participant
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Proportion of participant | 1

2. Secondary Outcome: Participants With Adverse Event by Grade
Description: Number participants with any adverse events by grade, up to 4 weeks after the final burosumab dose, was assessed using the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental ADL.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
  Grade 4 Life-threatening consequences; urgent intervention indicated.
  Grade 5 Death related to AE.
Time Frame: 48 weeks for adult participants; 50 weeks for pediatric participants
Population: Modified intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Participants
  Grade 1 | 9
  Grade 2 | 6
  Grade 3 | 1
  Grade 4 | 0
  Grade 5 | 0

3. Secondary Outcome: Participants With Related Adverse Event
Description: Participants with related adverse events up to 4 weeks after the final burosumab dose (48 weeks for adult subjects, 50 weeks for pediatric subjects). Adverse event was assessed using the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0. Related adverse event means that there are available evidence that suggests that there is a reasonable possibility that the study drug caused the adverse event.
Time Frame: 48 weeks for adult participants; 50 weeks for pediatric participants
Population: Modified intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Participants | 8

4. Secondary Outcome: Proportion of Participants With Serum Phosphate Levels Within the Target Range at Week 24
Description: The proportion of participants who achieved serum phosphate levels within the target range (Z-score -1 to +2) at week 24. Analysis was done by dividing the number of number of participants who achieved serum level by the number of participants analyzed.
Time Frame: Week 24
Population: Modified intent to treat population
Measure: Number; unit: Proportion of participants
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Proportion of participants | 0.92

5. Secondary Outcome: Proportion of Participants With Serum Phosphate Levels Above the Target Range (Z-score >+2)
Description: The proportion of participants who achieved serum phosphate levels above the target range (Z-score >+2) at any timepoint between baseline and week 48. Analysis was done by dividing the number of number of participants who achieved serum level above the target range by the number of participants analyzed.
Time Frame: Between baseline and week 48
Population: Modified intent to treat population
Measure: Number; unit: Proportion of participants
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Proportion of participants | 0.5

6. Secondary Outcome: Change in Serum Phosphate Level
Description: Change in serum phosphate level from baseline to week 48. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
mg/dL | 1.5 [0.8 to 2.2]

7. Secondary Outcome: Percent Change in Serum Phosphate Level
Description: Percent change in serum phosphate level from baseline to week 48. Measurements were taken at baseline and week 48. Analysis was done as percent change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: Percentage of change
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Percentage of change | 55.5 [29 to 106]

8. Secondary Outcome: Change in Serum 1,25-dihydroxyvitamin D Level
Description: Change in serum 1,25-dihydroxyvitamin D level from baseline to week 48. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
ng/mL | 7.5 [-19 to 57]

9. Secondary Outcome: Percent Change in Serum 1,25-dihydroxyvitamin D Level
Description: Percent change in serum 1,25-dihydroxyvitamin D level from baseline to 48 weeks. Measurements were taken at baseline and week 48. Analysis was done as percent change in median value between baseline and week 48. Change = 48 weeks minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: Percentage of change
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Percentage of change | 29.3 [-0.4 to 950]

10. Secondary Outcome: Change in Serum Ratio of Renal Tubular Maximum Reabsorption Rate of Phosphate to Glomerular Filtration Rate (TmP/GFR)
Description: Change in serum ratio of renal tubular maximum reabsorption rate of phosphate to glomerular filtration rate (TmP/GFR) from baseline to week 48. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
mmol/L | 0.51 [0.29 to 1.15]

11. Secondary Outcome: Percent Change in Serum Ratio of Renal Tubular Maximum Reabsorption Rate of Phosphate to Glomerular Filtration Rate (TmP/GFR)
Description: Percent change in serum ratio of renal tubular maximum reabsorption rate of phosphate to glomerular filtration rate (TmP/GFR) from baseline to week 48. Measurements were taken at baseline and week 48. Analysis was done as percent change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: Percentage of change
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Percentage of change | 68.05 [29.8 to 219]

12. Secondary Outcome: Change in Fibrous Dysplasia Lesion Activity Using Fluorine-18 Sodium Fluoride Positron Emission Tomography/Computed Tomography (18F-NaF PET/CT) Scan
Description: Change in fibrous dysplasia lesion activity using Fluorine-18 Sodium Fluoride Positron Emission Tomography/Computed Tomography (18F-NaF PET/CT) scan from baseline to week 48. 18F-NaF PET/CT scan was done at baseline and week 48 and total lesion activity units were calculated from each scan. Change in lesion activity was compared between timepoints, baseline and week 48. Change = 48 weeks minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: Total lesion activity units
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Total lesion activity units | 8.4 [-143 to 1518]

13. Secondary Outcome: Change in Serum Procollagen 1 N-terminal Propeptide (P1NP) Level
Description: Change in serum procollagen 1 N-terminal propeptide (P1NP) level from baseline to week 48. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: mcg/L
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
mcg/L | 8.5 [-611 to 1679]

14. Secondary Outcome: Percent Change in Serum Procollagen 1 N-terminal Propeptide (P1NP) Level
Description: Percent change in serum procollagen 1 N-terminal propeptide (P1NP) level from baseline to week 48. Measurements were taken at baseline and week 48. Analysis was done as percent change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: Percentage of change
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Percentage of change | 12.45 [-36.3 to 345]

15. Secondary Outcome: Change in Serum Beta Crosslaps C-telopeptides (CTX) Level
Description: Change in serum beta crosslaps C-telopeptides (CTX) level from baseline to week 48. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
pg/mL | 0.515 [0.29 to 1.15]

16. Secondary Outcome: Percent Change in Serum Beta Crosslaps C-telopeptides (CTX) Level
Description: Percent change in serum beta crosslaps C-telopeptides (CTX) level from baseline to week 48. Measurements were taken at baseline and week 48. Analysis was done as percent change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: Percentage of change
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Percentage of change | 1.69 [-34.6 to 138]

17. Secondary Outcome: Change in Serum Osteocalcin Level
Description: Change in serum osteocalcin level from baseline to week 48. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
ng/mL | 21.95 [-79.7 to 1184]

18. Secondary Outcome: Percent Change in Serum Osteocalcin Level
Description: Percent change in serum osteocalcin level from baseline to week 48. Measurements were taken at baseline and week 48. Analysis was done as percent change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: Percentage of change
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Percentage of change | 24.9 [-35 to 446]

19. Secondary Outcome: Change in Serum Alkaline Phosphatase Level
Description: Change in serum alkaline phosphatase level from baseline to week 48. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: U/L
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 8
U/L | -531.5 [-1493 to -147]

20. Secondary Outcome: Percent Change in Serum Alkaline Phosphatase Level
Description: Percent change in serum alkaline phosphatase level from baseline to week 48. Measurements were taken at baseline and week 48. Analysis was done as percent change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: Percentage of change
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 8
Percentage of change | -48.3 [-62.5 to -33.1]

21. Secondary Outcome: Change in Fibrous Dysplasia Lesion Cellularity
Description: Change in fibrous dysplasia lesion cellularity was assessed by minimally invasive bone biopsies at baseline and week 48 in only adult participants with capacity to consent to procedure. Bone biopsies assessed the count of cell density. Analysis was done as change in median cell density value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: Fibrosis nuclei/mcm^2
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 4
Fibrosis nuclei/mcm^2 | -0.0001163 [-0.001003 to 0.0001152]

22. Secondary Outcome: Change in Muscle Strength Using the Manual Muscle Test Scale
Description: Muscle strength was assessed using the manual muscle test (MMT) scale. MMT is a clinical technique to assess the strength of individual muscles or muscle groups based on ability to move against gravity and resist applied external pressure on a 0-5 scale, with 0 (no contraction), 1 (trace), 2 (poor) (movement with gravity eliminated), 3 (fair) (movement against gravity), 4 (good) (movement against gravity with moderate resistance), and 5 (normal strength). Higher number indicates better muscle resistance and strength. Each muscle group was assessed at baseline and week 48. Analysis was done for each muscle as change between baseline and week 48 (week 48 - baseline).
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population; participants were excluded from the specific muscle strength analysis if unable to complete the individual muscle strength test.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Units on a scale
  NECK_FLEXORS_RIGHT | 0 [-1 to 1]
  NECK_FLEXORS_LEFT: number analyzed (Participants) | 10
  NECK_FLEXORS_LEFT | 0 [-1 to 1]
  GLUTEUS_MEDIUS_RIGHT | 0 [-2 to 1]
  GLUTEUS_MEDIUS_LEFT | 0 [-1 to 1]
  GLUTEUS_MAXIMUS_RIGHT: number analyzed (Participants) | 11
  GLUTEUS_MAXIMUS_RIGHT | 0 [-1 to 1]
  GLUTEUS_MAXIMUS_LEFT: number analyzed (Participants) | 11
  GLUTEUS_MAXIMUS_LEFT | 0 [-3 to 1]
  HAMSTRINGS_RIGHT: number analyzed (Participants) | 11
  HAMSTRINGS_RIGHT | 0 [-1 to 1]
  HAMSTRINGS_LEFT: number analyzed (Participants) | 11
  HAMSTRINGS_LEFT | 0 [-1 to 1]
  ANKLE_PLANTAR_FLEXORS_RIGHT: number analyzed (Participants) | 10
  ANKLE_PLANTAR_FLEXORS_RIGHT | 0 [-1 to 1]
  ANKLE_PLANTAR_FLEXORS_LEFT: number analyzed (Participants) | 10
  ANKLE_PLANTAR_FLEXORS_LEFT | 0 [0 to 1]
  NECK_EXTENSORS_RIGHT | 0 [0 to 0]
  NECK_EXTENSORS_LEFT: number analyzed (Participants) | 11
  NECK_EXTENSORS_LEFT | 0 [0 to 0]
  TRAPEZIUS_RIGHT | 0 [0 to 1]
  TRAPEZIUS_LEFT | 0 [0 to 1]
  DELTOID_RIGHT | 0 [0 to 1]
  DELTOID_LEFT | 0 [0 to 1]
  BICEPS_BRACHII_RIGHT | 0 [0 to 1]
  BICEPS_BRACHII_LEFT | 0 [0 to 2]
  ILIOPSOAS_RIGHT: number analyzed (Participants) | 11
  ILIOPSOAS_RIGHT | 0 [-3 to 1]
  ILIOPSOAS_LEFT: number analyzed (Participants) | 11
  ILIOPSOAS_LEFT | 0 [-3 to 3]
  QUADRICEPS_RIGHT | 0 [-2 to 1]
  QUADRICEPS_LEFT | 0 [-2 to 1]
  WRIST_FLEXORS_RIGHT | 0 [0 to 1]
  WRIST_FLEXORS_LEFT | 0 [0 to 2]
  WRIST_EXTENSORS_RIGHT | 0 [0 to 1]
  WRIST_EXTENSORS_LEFT | 0 [0 to 2]
  HALLUCIS_LONGUS_EXTENSOR_RIGHT | 0 [0 to 1]
  HALLUCIS_LONGUS_EXTENSOR_LEFT | 0 [0 to 1]
  ANKLE_DORSIFLEX_RIGHT | 0 [0 to 1]
  ANKLE_DORSIFLEX_LEFT | 0 [0 to 1]

23. Secondary Outcome: Change in Muscle Range-of-motion
Description: Muscle range-of-motion was measured as the degree of movement of muscles. Assessment was done at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: as for outcome 22
Measure: Median (Full Range); unit: Degrees
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Degrees
  SHOULDER_ABDUCTION_RIGHT | 0 [0 to 17]
  SHOULDER_ABDUCTION_LEFT | 0 [-21 to 9]
  SHOULDER_INTERNAL_ROTATION_RIGHT | 0 [0 to 38]
  SHOULDER_INTERNAL_ROTATION_LEFT | 0 [-22 to 45]
  SHOULDER_EXTERNAL_ROTATION_RIGHT | 0 [-15 to 39]
  SHOULDER_EXTERNAL_ROTATION_LEFT | 0 [0 to 12]
  ELBOW_FLEXION_RIGHT | -5 [-17 to 10]
  ELBOW_FLEXION_LEFT | -6 [-19 to 8]
  ELBOW_EXTENSION_RIGHT | -0.5 [-9 to 1]
  ELBOW_EXTENSION_LEFT | -1 [-7 to 3]
  WRIST_FLEXION_RIGHT | 18 [-15 to 27]
  WRIST_FLEXION_LEFT | 21 [-19 to 105]
  WRIST_EXTENSION_RIGHT | 12.5 [-20 to 28]
  WRIST_EXTENSION_LEFT | 5 [-15 to 87]
  HIP_FLEXION_RIGHT | 4 [-20 to 19]
  HIP_FLEXION_LEFT | -4 [-24 to 34]
  HIP_EXTENSION_RIGHT: number analyzed (Participants) | 11
  HIP_EXTENSION_RIGHT | 0 [-10 to 10]
  HIP_EXTENSION_LEFT | 2.5 [-13 to 15]
  HIP_EXTENSION_ROTATION_RIGHT | 0 [-25 to 42]
  HIP_EXTENSION_ROTATION_LEFT | -4.5 [-28 to 32]
  HIP_INTERNAL_ROTATION_RIGHT | 3.5 [-17 to 39]
  HIP_INTERNAL_ROTATION_LEFT | -4 [-11 to 38]
  HIP_ABDUCTION_RIGHT | 8.5 [-30 to 30]
  HIP_ABDUCTION_LEFT | 11 [-57 to 41]
  KNEE_FLEXION_RIGHT | -3.5 [-19 to 15]
  KNEE_FLEXION_LEFT | -5 [-25 to 6]
  KNEE_EXTENSION_RIGHT | 0 [-15 to 5]
  KNEE_EXTENSION_LEFT | 0 [-16 to 24]
  ANKLE_PLANTARFLEXION_RIGHT | -2 [-18 to 17]
  ANKLE_PLANTARFLEXION_LEFT | 8 [-14 to 29]
  ANKLE_DORSIFLEXION_RIGHT | -0.5 [-6 to 9]
  ANKLE_DORSIFLEXION_LEFT | -0.5 [-10 to 24]

24. Secondary Outcome: Change in Walking Speed Measured by the 9-minute Walk Test (9MWT)
Description: Change in walking speed was measured by the 9-minute walk test from baseline to week 48. The 9-minute walk test (9MWT) is a measure of physical capacity and participants are instructed to run or walk over a time period of nine minutes. The 9-minute walk test distance (9MWD) is the total distance walked in meters during the 9MWT and greater distance walked means better physical capacity. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population; analysis excludes non-ambulatory participants.
Measure: Median (Full Range); unit: Meters
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 5
Meters | 3 [-369 to 570]

25. Secondary Outcome: Change in Quality of Life Measured by the 36-Item Short Form Health Survey (SF-36) Score
Description: The change in quality of life for the adult participants was assessed using the Short Form Health Survey (SF-36). SF-36 is a 36-item patient-reported survey of patient health status that consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. The higher the score, the less disability. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 5
Units on a scale | 5 [-10 to 25]

26. Secondary Outcome: Change in Health-related Quality of Life Measured by the 10-Item Short Form Health Survey (SF-10) - Physical Summary Score (PHS)
Description: The change in quality of life for the pediatric participants was assessed using the Short-Form Health Survey-10 (SF-10). The Short-Form Health Survey (SF-10) is a 10-item parent-completed questionnaire that covers a wide range of domains affecting a child's functional health and well-being. The SF-10 is scored to produce two norm-based summary scores: a Physical Summary Score (PHS) and a Psychosocial Summary Score (PSS), each with a mean of 50 and a standard deviation of 10. Analysis was based on the PHS. The PHS scale is directly transformed into a 0-100 scale. The higher the score, the less disability. Measurements were taken for the Physical Summary Score (PHS) at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 7
Units on a scale | 16.63 [-19.78 to 39.28]

27. Secondary Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS) Score (Pediatric and Parent Proxy Version 1.0) - Pain Intensity Domain
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity (Pediatric and Parent Proxy version 1.0) domain measures pain intensity in children, with pediatric self-report versions for ages 8-17 and parent proxy-report versions for children aged 5-17. This measure uses a standard scale to assess the level of pain over the past seven days, and for the current moment, providing a quantitative score that reflects the severity of the pain. The scale consist of three items with each scored on a 5-point Likert scale, 1-5 with lowest score of 3 and highest of 15. The raw score is converted to a T-score with a mean of 50 and standard deviation of 10. Higher scores indicates greater pain intensity. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: T-Score
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 7
T-Score | -1 [-7 to 0]

28. Secondary Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS) Score (Adult Version 2.0) - Pain Intensity Domain
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity (Adult version 2.0) - Pain Intensity domain is a universal, self-report measure of how much pain a person is experiencing. This measure uses a standard scale to assess the level of pain over the past seven days, and for the current moment, providing a quantitative score that reflects the severity of the pain. The scale consist of three items with each scored on a 5-point Likert scale, 1-5 with lowest score of 3 and highest of 15. The raw score is converted to a T-score with a mean of 50 and standard deviation of 10. Higher scores indicates greater pain intensity. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: T-Score
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 5
T-Score | 5.8 [-7.3 to 19.8]

29. Secondary Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS) Score (Pediatric and Parent Proxy Version 2.0) - Pain Inference Domain
Description: The Patient Reported Outcome Measurement Information System (PROMIS) (Pediatric and Parent Proxy version 2.0) - Pain Inference Domain assesses how pain impacts daily life, sleep, and enjoyment in children, with the Pediatric version being self-reported by children aged 8-17 and the Parent Proxy version completed by a parent or guardian for their child aged 5-17. This measure uses a standard scale to assess the level of pain interference over the past seven days, and for the current moment, providing a quantitative score that reflects the severity of the pain interference. Each item is rated on a 5-point scale (1-5). The scores are then summed and converted into a T-score, with a mean of 50 and standard deviation of 10. Higher scores indicate greater pain interference. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: T-Score
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 7
T-Score | 0 [-27 to 1.6]

30. Secondary Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS) Score (Adult Version 1.1) - Pain Inference Domain
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) (Adult version 1.1) - Pain Inference scale assesses the impact of pain on social, physical, cognitive, emotional, and recreational activities, as well as sleep and life enjoyment. The scale consists of 12 items and each item is rated on a 5-point scale (1-5). The scores are then summed and converted into a T-score, with a mean of 50 and standard deviation of 10. Higher scores indicate greater pain interference. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: T-Score
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 5
T-Score | 0.2 [-0.2 to 1.6]

31. Secondary Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS) Score (Pediatric and Parent Proxy Version 2.0) - Mobility Lower Extremity Domain
Description: The Patient Reported Outcome Measurement Information System (PROMIS) (Pediatric and Parent Proxy version 2.0) Mobility Lower Extremity domain assesses self-perceived mobility in children, with the Pediatric version being self-reported by children aged 8-17 and the Parent Proxy version completed by a parent or guardian for their child aged 5-17. This measure uses a standard scale to assess lower extremity mobility by asking about activities such as getting up from a chair or running over the past seven days. Each item is rated on a 5-point scale (1-5). The scores are then summed and converted into a T-score, with a mean of 50 and standard deviation of 10. Higher scores indicate greater mobility. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: T-Score
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 7
T-Score | 11.1 [-4.3 to 21.3]

32. Secondary Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS) Score (Adult Version 2.0) - Mobility Lower Extremity Domain
Description: The Patient Reported Outcome Measurement Information System (PROMIS) (Adult version 2.0) Mobility Lower Extremity Domain assesses an adult's self-perceived ability to perform physical tasks related to mobility and lower extremity function, such as getting out of a chair or walking. This measure uses a standard scale to assess lower extremity mobility by asking about mobility activities over the past seven days. Each item is rated on a 5-point scale (1-5). The scores are then summed and converted into a T-score, with a mean of 50 and standard deviation of 10. Higher scores indicate greater mobility. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Median (Full Range); unit: T-Score
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 5
T-Score | 0.5 [-8.4 to 6.3]

33. Secondary Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS) Score (Pediatric and Parent Proxy Version 2.0) - Fatigue Domain
Description: The Patient Reported Outcome Measurement Information System (PROMIS) (Pediatric and Parent Proxy version 2.0) Fatigue domain assess the level and impact of fatigue in children and adolescents, with the Pediatric version being self-reported by children aged 8-17 and the Parent Proxy version completed by a parent or guardian for their child aged 5-17. This measure uses a standard scale to assess the level of fatigue over the past seven days. Each item is rated on a 5-point scale (1-5). The scores are then summed and converted into a T-score, with a mean of 50 and standard deviation of 10 based on a US general population. Higher scores indicate worsening fatigue. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48
Population: Modified intent to treat population
Measure: Median (Full Range); unit: T-Score
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 7
T-Score | -6.5 [-28.3 to 4]

34. Secondary Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS) - Short Form - Fatigue 13a (Adult FACIT 13a v1.0)
Description: The Patient Reported Outcome Measurement Information System (PROMIS) Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Scale is a 13-item patient-reported outcome (PRO) questionnaire that captures the individual's subjective experience of their fatigue. The fatigue domain is scored on a 5-point Likert scale and converted into standardized T-scores with a mean of 50 and a standard deviation of 10 based on a US general population. Higher score indicates less fatigue. Measurements were taken at baseline and week 48. Analysis was done as change in median value between baseline and week 48. Change = week 48 minus baseline.
Time Frame: Week 48
Population: Modified intent to treat population
Measure: Median (Full Range); unit: T-Score
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 5
T-Score | 0 [-9.6 to 16]

35. Secondary Outcome: Proportion of Participants With Change in Activities of Daily Living (ADL) Questions
Description: Proportion of participants with change in activities of daily living (ADL) questions from baseline to week 48 was assessed using a study developed questionnaire. Participants and/or caregivers were asked to provide a list of three activities of daily living that were affected by fibrous dysplasia skeletal features at home or school/work (e.g., mobility, climbing stairs, dressing, playing with peers, catching a bus, etc.) and to rate the extent of impact upon their activity level using one of the option:
  * Very Much Improved
  * Much Improved
  * Minimally Improved
  * No Change
  * Minimally Worse
  * Much Worse
  * Very Much Worse
  These activities were assessed at baseline, then reassessed at Week 24 and Week 48. Analysis was done as proportion of participants reporting "much improved" or "very much improved" in Activities of Daily Living Questions. Change = Week 48 minus baseline.
Time Frame: Week 48 minus baseline
Population: Modified intent to treat population
Measure: Number; unit: Proportion of participants
Arm/Group | Treatment With Burosumab
Number analyzed (Participants) | 12
Proportion of participants | 0.67

ADVERSE EVENTS:
Time Frame: 48 weeks for adult participants; 50 weeks for pediatric participants
Arm/Group | Treatment With Burosumab
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Burosumab (N=12)
Appendicitis (Gastrointestinal disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hospitalisation (Surgical and medical procedures) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Burosumab (N=12)
Diarrhoea (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Injection site reaction (General disorders) | 3
Bacterial infection (Infections and infestations) | 1
Corona virus infection (Infections and infestations) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin infection (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT05509595/Prot_SAP_000.pdf